CLINICAL TRIAL: NCT03118349
Title: Phase I, Open-Label, Multi-Center, Dose Escalation With Expansion Trial of 177Lu Human Monoclonal Antibody 5B1 (MVT-1075) in Combination With a Blocking Dose of MVT-5873 as Radioimmunotherapy in Relapse/Refractory Subjects With Pancreatic Cancer or Other CA19-9 Positive Malignancies
Brief Title: Study of 177Lu Human Monoclonal Antibody 5B1 (MVT-1075) in Combination With a Blocking Dose of MVT-5873 as Radioimmunotherapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: BioNTech Research & Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: BioNTech SE (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MV-0916-CP-001.01
Record Dates: First submitted 2017-03-23; First posted 2017-04-18 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Pancreatic Carcinoma; Tumors That Express CA 19-9
Keywords: CA19-9 Positive Malignancies
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Escalation Cohorts (Experimental): MVT-5873 blocking dose and MVT-1075 dose escalation; Initial to maximum tolerated dose
  Interventions: Drug: MVT-1075; Drug: MVT-5873
- Expansion Cohort - no subjects enrolled (Experimental): MVT-5873 blocking dose and MVT-1075 Maximum tolerated dose
  Interventions: Drug: MVT-1075; Drug: MVT-5873

INTERVENTIONS:
Drug: MVT-1075 — MVT-1075 administered in two fractions, with each administration of MVT-1075 preceded by blocking dose of MVT-5873.
  Other Names: 177Lu-CHX-A"-DTPA-HuMab-5B1
Drug: MVT-5873 — MVT-5873 administered intravenously as a non-radioactive blocking agent prior to administration of MVT-1075.
  Other Names: HuMab-5B1

SUMMARY:
Open label, nonrandomized, dose-escalation with cohort expansion study of MVT-5873/MVT-1075 in subjects with previously treated, Carbohydrate Antigen 19-9 (CA19-9) positive malignancies (e.g., pancreatic adenocarcinoma).

DETAILED DESCRIPTION:
Open label, nonrandomized, dose escalation study of MVT-5873/MVT-1075 to evaluate safety, dosimetry, determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D), and define the pharmacokinetics of MVT-1075. The population consisted of subjects with CA19-9 positive malignancies (i.e., predominately pancreatic adenocarcinoma) who may benefit from a CA19-9-based radioimmunotherapy.

The study utilized a 3+3 study design to identify the MTD. The RP2D was planned to be no higher than the MTD. An expansion group was planned to receive MVT-5873/MVT-1075 at the RP2D in order to obtain initial estimates of response and additional information on safety.

ELIGIBILITY:
Inclusion Criteria:

1. Signed, informed consent
2. Age 18 or more years
3. Histologically or cytologically confirmed, previously treated, locally-advanced or metastatic pancreatic ductal adenocarcinoma (PDAC) or other CA19-9 positive malignancies
4. Prior treatment with (or intolerance to) at least one standard systemic regimen for the patient's respective tumor
5. Evidence of tumor expression of CA19-9 based on immunohistochemistry performed on tumor samples or elevated serum levels (≥1.5 x upper limits of normal [ULN]) of CA19-9 considered secondary to tumor
6. Evaluable or measurable disease based on RECIST 1.1
7. Recovered from any prior treatment related toxicity to at least Grade 1 with exception of Grade 2 alopecia or other Grade 2 toxicity with prior approval of the Medical Monitor
8. If previously exposed to irradiation, the combined prior and anticipated exposure for Cycle 1 is not expected to exceed organ exposure limits outlined in the study protocol
9. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, or Karnofsky performance status (KPS) of 100% to 80%
10. Adequate hematologic, renal and hepatic laboratory parameters
11. Willingness to participate in collection of pharmacokinetic samples
12. Willingness to use adequate contraception throughout study and for a period of 3 months after last dose of MVT-5873 or MVT-1075 (whichever is later)

Exclusion Criteria:

1. Brain metastases unless previously treated and well controlled for at least 3 months
2. Any tumor mass greater than 10 cm in longest diameter
3. Other known active cancer(s) likely to require treatment in the next two years
4. Active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy
5. Prior radiation therapy encompassing more than 25% of the skeleton or prior treatment with 89Strontium or 153Samarium
6. Fewer than 28 days from prior anticancer therapy including chemotherapy, hormonal, investigational, and/or biological therapies and irradiation except for:

   1. Ongoing hormonal therapy administered for control of cancer (e.g., breast cancer, prostate cancer), which may be continued throughout the study
   2. MVT-5873 and MVT-2163 administered as part of a different protocol
7. Major surgery other than diagnostic surgery within 28 days of Study Day 1
8. History of anaphylactic reaction to human, or humanized, antibody
9. Pregnant or currently breast-feeding
10. Known to be positive for human immunodeficiency virus (HIV), Hepatitis B, or Hepatitis C
11. Psychiatric illness/social situations that would interfere with compliance with study requirements
12. Significant cardiovascular risk including, but not limited to, recent (within 4 weeks) coronary stenting or myocardial infarction within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-04-11 (Actual); Study Completion 2018-04-11 (Actual)

PRIMARY OUTCOMES:
The MTD of MVT-5873/MVT-1075 | Through study completion. Estimated at one year
  The MTD of MVT-5873/MVT-1075 is the highest dose of MVT-1075 at which fewer than 33% subjects experience a dose limiting toxicity
Occurrence of graded adverse events (AEs) in each subject | Through study completion. Estimated at one year
  Occurrence of graded AEs in each subject

SECONDARY OUTCOMES:
Specific organ distribution of MVT-1075 as assessed with planar gamma camera | Through study completion. Estimated at one year
  Specific organ distribution of MVT-1075 as assessed with planar gamma camera
Specific organ distribution of MVT-1075 as assessed with single-photon emission computed tomography (SPECT) imaging | Through study completion. Estimated at one year
  Specific organ distribution of MVT-1075 as assessed with SPECT imaging
A RP2D of MVT-5873/MVT-1075 | Through study completion. Estimated at one year.
  Previously determined MTD; Overall assessment of safety as determined by Safety Committee
Evaluate the tumor response rate to MVT-5873/MVT-1075 at the RP2D | Through study completion. Estimated at one year.
  Response categories as assessed by Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST v1.1)
Evaluate duration of response of MVT-5873/MVT-1075 | Through study completion. Estimated at one year.
  Time from first onset of response to progression or death
Evaluate formation of anti-drug antibodies (ADA) | On Day 1, Day 15 and End of Treatment Visit only of each cycle for up to 4 cycles. (each cycle is 57 days)
  Presence or absence of ADA as assessed by assay to be developed
Cmax | Measured on Day 1 Prior to MVT-1075 dose and again 15 min. 30 min. 60 min. 120 min. post MVT-1075 dose. On Day 3, Day 8, Day 15 Prior and 15 min Post MVT-1075 dose. Anytime on Day 22 and Day 29. During cycle 1 and 2 only (each cycle is 57 days).
  The peak plasma concentration of the drug after administration
Cmin | Measured on Day 1 Prior to MVT-1075 dose and again 15 min. 30 min. 60 min. 120 min. post MVT-1075 dose. On Day 3, Day 8, Day 15 Prior and 15 min Post MVT-1075 dose. Anytime on Day 22 and Day 29. During cycle 1 and 2 only (each cycle is 57 days).
  Measure the lowest concentration that the drug reaches before the next dose is administered.
Tmax | Measured on Day 1 Prior to MVT-1075 dose and again 15 min. 30 min. 60 min. 120 min. post MVT-1075 dose. On Day 3, Day 8, Day 15 Prior and 15 min Post MVT-1075 dose. Anytime on Day 22 and Day 29. During cycle 1 and 2 only (each cycle is 57 days).
  Time to reach the study drug
Vd | Measured on Day 1 Prior to MVT-1075 dose and again 15 min. 30 min. 60 min. 120 min. post MVT-1075 dose. On Day 3, Day 8, Day 15 Prior and 15 min Post MVT-1075 dose. Anytime on Day 22 and Day 29. During cycle 1 and 2 only (each cycle is 57 days).
  Volume of distribution
t1/2 | Measured on Day 1 Prior to MVT-1075 dose and again 15 min. 30 min. 60 min. 120 min. post MVT-1075 dose. On Day 3, Day 8, Day 15 Prior and 15 min Post MVT-1075 dose. Anytime on Day 22 and Day 29. During cycle 1 and 2 only (each cycle is 57 days).
  Half-life of Elimination
AUC | Measured on Day 1 Prior to MVT-1075 dose and again 15 min. 30 min. 60 min. 120 min. post MVT-1075 dose. On Day 3, Day 8, Day 15 Prior and 15 min Post MVT-1075 dose. Anytime on Day 22 and Day 29. During cycle 1 and 2 only (each cycle is 57 days).
  Area under the plasma concentration time curve
Cl | Measured on Day 1 Prior to MVT-1075 dose and again 15 min. 30 min. 60 min. 120 min. post MVT-1075 dose. On Day 3, Day 8, Day 15 Prior and 15 min Post MVT-1075 dose. Anytime on Day 22 and Day 29. During cycle 1 and 2 only (each cycle is 57 days).
  Clearance of study drug

OTHER OUTCOMES:
Evaluate the relationship between circulating CA19-9 levels and tumor response | Through study completion. Estimated at one year.
  Periodic assessment of CA19-9 expression
Evaluate the relationship between circulating CA19-9 levels and MVT-1075 pharmacokinetics | Through study completion. Estimated at one year.
  Periodic assessments pre and post MVT-1075

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (2):
- United States (2):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - MSKCC, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tully KM, Tendler S, Carter LM, Sharma SK, Samuels ZV, Mandleywala K, Korsen JA, Delos Reyes AM, Piersigilli A, Travis WD, Sen T, Pillarsetty N, Poirier JT, Rudin CM, Lewis JS. Radioimmunotherapy Targeting Delta-like Ligand 3 in Small Cell Lung Cancer Exhibits Antitumor Efficacy with Low Toxicity. Clin Cancer Res. 2022 Apr 1;28(7):1391-1401. doi: 10.1158/1078-0432.CCR-21-1533. PMID 35046060